CLINICAL TRIAL: NCT01495754
Title: The Effect of Different Amounts of Coffee on Dietary Intake, Appetite-related Feeling, Appetite Hormones, Glucose Metabolism and Inflammatory Markers of Normal Weight and Overweight/Obese Individuals
Brief Title: Effects of Different Coffee Amounts on Energy Intake, Appetite, Glucose Metabolism and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, M. Yannakoulia, Assistant Professor, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CofSt3
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Obesity; Inflammation
Keywords: coffee; overweight/obese; appetite; energy intake; inflammation; glucose metabolism; randomized controlled trial
MeSH Terms: conditions — Obesity; Inflammation; Overweight | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- coffee3 (Experimental)
  Interventions: Other: coffee
- coffee6 (Experimental)
  Interventions: Other: coffee
- water (Placebo Comparator)
  Interventions: Other: coffee

INTERVENTIONS:
Other: coffee — Comparison of different amounts of coffee

SUMMARY:
The purpose of the study is to investigate whether different doses of caffeinated coffee consumption has acute effects on subjective appetite feelings, energy intake and biochemical markers related to appetite, inflammation and glucose metabolism compared to water consumption in normal weight and overweight/obese participants.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy
* habitual coffee drinkers (>= 1cup of coffee/day)

Exclusion Criteria:

* smokers
* restrained eaters (as this was evaluated using the Dutch Eating Behaviour Questionnaire)
* those who reported slimming or any other dietary regime
* athletes
* participants with a known diagnosis of either hypertension, diabetes, impaired glucose tolerance or a fasting blood glucose concentration above 125 mg/dl
* subjects on medication for hypertension or on medication known to alter glucose metabolism
* subjects who were on medication that may have an impact on appetite and sensory functioning or who reported a metabolic or
* endocrine disease,
* gastrointestinal disorders,
* a history of medical or surgical events that may have affected the study outcomes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
energy intake ad libitum | 180 min after breakfast/drink consumption
total energy intake | One day
appetite feelings | fasting (-15 min)
appetite feelings | immediately after breakfast/drink consumption (0 min)
appetite feelings | 15 min after breakfast/drink consumption
appetite feelings | 30 min after breakfast/drink consumption
appetite feelings | 60 min after breakfast/drink consumption
appetite feelings | 90 min after breakfast/drink consumption
appetite feelings | 120 min after breakfast/drink consumption
appetite feelings | 150 min after breakfast/drink consumption
appetite feelings | 180 min after breakfast/drink consumption
appetite hormones | fasting (-15 min)
appetite hormones | immediately after breakfast/drink consumption (0 min)
appetite hormones | 15 min after breakfast/drink consumption
appetite hormones | 30 min after breakfast/drink consumption
appetite hormones | 60 min after breakfast/drink consumption
appetite hormones | 90 min after breakfast/drink consumption
appetite hormones | 120 min after breakfast/drink consumption
appetite hormones | 150 min after breakfast/drink consumption
appetite hormones | 180 min after breakfast/drink consumption
markers of inflammation | fasting (-15 min)
markers of inflammation | immediately after breakfast/drink consumption (0 min)
markers of inflammation | 15 min after breakfast/drink consumption
markers of inflammation | 30 min after breakfast/drink consumption
markers of inflammation | 60 min after breakfast/drink consumption
markers of inflammation | 90 min after breakfast/drink consumption
markers of inflammation | 120 min after breakfast/drink consumption
markers of inflammation | 150 min after breakfast/drink consumption
markers of inflammation | 180 min after breakfast/drink consumption
markers of glucose metabolism | fasting (-15 min)
markers of glucose metabolism | immediately after breakfast/drink consumption (0 min)
markers of glucose metabolism | 15 min after breakfast/drink consumption
markers of glucose metabolism | 30 min after breakfast/drink consumption
markers of glucose metabolism | 60 min after breakfast/drink consumption
markers of glucose metabolism | 90 min after breakfast/drink consumption
markers of glucose metabolism | 120 min after breakfast/drink consumption
markers of glucose metabolism | 150 min after breakfast/drink consumption
markers of glucose metabolism | 180 min after breakfast/drink consumption

SECONDARY OUTCOMES:
% carbohydrates ad libitum | 180 min after breakfast/drink consumption
% carbohydrates total day | One day
% protein ad libitum | 180 min after breakfast/drink consumption
% protein total day | One day
% fat | 180 min after breakfast/drink consumption
% fat total day | One day

CONTACTS AND LOCATIONS:
Overall Officials: Mary Yannakoulia, PhD, Principal Investigator — Harokopio University
Locations (1):
- Metabolic Unit of the Department of Nutrition and Dietetics, Harokopio University, Athens, Greece

REFERENCES:
- [Background] Gavrieli A, Yannakoulia M, Fragopoulou E, Margaritopoulos D, Chamberland JP, Kaisari P, Kavouras SA, Mantzoros CS. Caffeinated coffee does not acutely affect energy intake, appetite, or inflammation but prevents serum cortisol concentrations from falling in healthy men. J Nutr. 2011 Apr 1;141(4):703-7. doi: 10.3945/jn.110.137323. Epub 2011 Feb 23. PMID 21346100
- [Derived] Perakakis N, Kokkinos A, Angelidi AM, Tsilingiris D, Gavrieli A, Yannakoulia M, Tentolouris N, Mantzoros CS. Circulating levels of five proglucagon-derived peptides in response to intravenous or oral glucose or lipids and to a mixed-meal in subjects with normal weight, overweight, and obesity. Clin Nutr. 2022 Sep;41(9):1969-1976. doi: 10.1016/j.clnu.2022.07.001. Epub 2022 Jul 19. PMID 35961260
- [Derived] Gavrieli A, Fragopoulou E, Mantzoros CS, Yannakoulia M. Gender and body mass index modify the effect of increasing amounts of caffeinated coffee on postprandial glucose and insulin concentrations; a randomized, controlled, clinical trial. Metabolism. 2013 Aug;62(8):1099-106. doi: 10.1016/j.metabol.2013.02.003. Epub 2013 Mar 15. PMID 23498899